CLINICAL TRIAL: NCT03716362
Title: Neonatal Hearing Screening at Neonatal Intensive Care Unit of Assiut University Hospital
Brief Title: Neonatal Hearing Screening at Neonatal Intensive Care Unit
Status: Withdrawn | Type: Observational
Why Stopped: no participant
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Other Study IDs: NHS
Record Dates: First submitted 2018-10-21; First posted 2018-10-23 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates who will be admitted at Neonatal Intensive Care Unite
  Interventions: Device: Otoacoustic emissions device

INTERVENTIONS:
Device: Otoacoustic emissions device — as a screening tool for Auditory brainstem response

SUMMARY:
Hearing loss is one of the most common congenital anomalies . It has been shown to be greater than that of most other diseases and syndromes (eg, phenylketonuria, sickle cell disease) screened at birth. Data from the newborn hearing-screening programs in Rhode Island, Colorado, and Texas showed that 2-4 of every 1000 neonates have hearing loss.

Early Intervention at or before 6 months of age allows a child with impaired hearing to develop normal speech and language, alongside his or her hearing peers and can prevent severe psychosocial, educational, and language impairment.

One of the most high risk population are neonates who spend time in the newborn intensive care unit , exposed to high frequency ventilation, hyperbilirubinemia, low birth-weight, and exposed to ototoxic medications.

Auditory brainstem response , otoacoustic emissions , and automated Auditory brainstem response testing have all been used in newborn hearing-screening programs. otoacoustic emissions are fast objective, efficient, and frequency-specific measurements of peripheral auditory sensitivity are used to assess response of the outer hair cells to acoustic stimuli. To measure otoacoustic emissions, a probe assembly is placed in the ear canal, tonal or click stimuli are delivered, and the otoacoustic emissions generated by the cochlea is measured with a microphone .

ELIGIBILITY:
Inclusion Criteria:

* Neonates of both sexes.
* Neonates with In utero infection such as cytomegalovirus, rubella, toxoplasmosis, or herpes.
* Neonatal indicators, specifically hyperbilirubinemia at a serum level requiring exchange transfusion.

Exclusion Criteria:

* neonates whose parent refuse to participate in the study.

Ages: 1 Week to 4 Weeks | Sex: All
Age Groups: Child
Study Population: This study will conduct on neonates who will be admitted at intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hearing loss in all neonates in Neonatal Intensive Care Unit | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided